CLINICAL TRIAL: NCT04350164
Title: Retrospective Chart Review of Children With Wiskott-Aldrich Syndrome Who Received Romiplostim in Treatment of Thrombocytopenia.
Brief Title: Romiplostim Treatment for Thrombocytopenia in Patients With Wiskott-Aldrich Syndrome.
Status: Completed | Type: Observational
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Other Study IDs: NCPHOI-2020-02
Record Dates: First submitted 2020-04-10; First posted 2020-04-16 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Wiskott-Aldrich Syndrome
MeSH Terms: conditions — Wiskott-Aldrich Syndrome | interventions — romiplostim

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- treatment: romiplostim once weekly subcutaneously at an initial dose of 8-9 µg/kg per week for at least 1 month to 1 year.
  Interventions: Drug: Romiplostim

INTERVENTIONS:
Drug: Romiplostim — romiplostim once weekly subcutaneously at an initial dose of 8-9 µg/kg per week for at least 1 month to 1 year.
  Other Names: Nplate

SUMMARY:
The rationale for this retrospective study is to evaluate the efficacy and safety of thrombopoietin-receptor agonist (TPO-RA) romiplostim for reducing thrombocytopenia and bleeding tendency in pediatric participants with genetically confirmed Wiskott-Aldrich syndrome (WAS).

DETAILED DESCRIPTION:
Thrombocytopenia is a life-threatening symptom in WAS patients. Subjects with WAS are at increased risk of debilitating and\ or life-threatening bleedings due to low platelet numbers. Hematopoietic stem cell transplantation is an effective treatment of WAS and all its symptoms yet requires time for donor search and is not widely utilized in cases with mild WAS with isolated thrombocytopenia. TPO-RAs have been used in individual WAS patients, wherein publications describing large WAS cohorts treated with TPO-RAs are lacking.

Based on the previous reports, WAS patients in our Center have been receiving treatment with TPO-RA romiplostim since 2012.

The aim of the study is to retrospective analyze patients' data in order to asses treatment efficacy and safety of romiplostim in WAS thrombocytopenia.

The study will collect and analyze information that is already in the patients' medical records. Information about clinical data (assessment of bleeding tendency with a modified World Health Organization (WHO) Bleeding Scale), laboratory values (such as clinical and biochemical analysis of blood) will be included.

Evaluation of the efficacy therapy was based on the results of physical examination, including bleeding events at the time of diagnosis and after 6-month TPO-RA was initiated and platelet response. A complete response was defined as a platelet count >100 x 109/L in the absence of bleeding symptoms, partial - 30 x 109/L higher than the patient's pretreatment baseline count to 100 x 109/L. Non-response was defined as not achieving a platelet count of > 30 x 109/L from the baseline count.

ELIGIBILITY:
Inclusion Criteria:

* Age under < 18 years
* Subject/legal representative has signed written informed consent. ?
* Subjects diagnosed with WAS based on genetic findings.
* Subjects with thrombocytopenia (platelet count of less than 70 x 109/L).
* Subjects with a history of bleeding.
* Subjects received treatment with romiplostim 8-9 µg /kg for at least 30 days
* Available records of the points of analysis

Exclusion Criteria:

• Patients, who do not meet the inclusion criteria.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients of the immunology department
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
The percentage of participants with overall platelet response (complete response + partial response) | 1 month (30 day +/- 14 days)
  A complete response defined as a platelet count >100 x 109/L, partial - 30 x 109/L higher than the patient's pretreatment baseline count to 100 x 109/L.

SECONDARY OUTCOMES:
Percentage of patients with a platelet response | until discontinuation, from at least one month to one year
Number of participants with bleeding events and severity of bleeding | until discontinuation, from at least one month to one year
  The incidence and severity of bleeding events evaluated with a modified World Health Organization (WHO) Bleeding Scale.
  (G1=Petechiae, epistaxis <30 min, G2=Mild blood loss, hematomas, epistaxis >30 min, melanotic stool G3=Gross blood loss, requiring blood transfusions, G4=Fatal bleeding).
Number of participants with adverse events | until discontinuation, from at least one month to one year

CONTACTS AND LOCATIONS:
Overall Officials: Anna Shcherbina, MD, PhD, Principal Investigator — National Research Center for Pediatric Hematology , Moscow, Russian Federation
Locations (1):
- Dmitry Rogachev National Research Center of Pediatric Hematology, Oncology and Immunology, Moscow, Russia